CLINICAL TRIAL: NCT01584284
Title: Phase I Trial Of Attenuated Vaccinia Virus (GL-ONC1) Delivered Intravenously With Concurrent Cisplatin and Radiotherapy in Patients With Locoregionally Advanced Head and Neck Carcinoma
Brief Title: Safety Study of Attenuated Vaccinia Virus (GL-ONC1)With Combination Therapy in Head & Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genelux Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-ONC1-005
Record Dates: First submitted 2012-04-22; First posted 2012-04-24 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Cancer of Head and Neck
Keywords: Genelux; Genelux Corporation; GL-ONC1; Vaccinia; Vaccinia Virus; Oncolytic virus; Oncolytic Virotherapy; Head and Neck Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Vaccinia; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: GL-ONC1 — A genetically-engineered vaccinia virus administered via intravenous infusion . Cohorts 1, 2, 3: Frequency: 1x in Week 1; Cohort 4: 1x again 1x in Week 2; Cohort 5: 1x Week 1, 1x Week 2, 1x Week 3, 1x Week 4.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of GL-ONC1 administered intravenously in combination with radiation therapy and cisplatin (CDDP)in patients with locoregionally advanced head and neck cancer.

DETAILED DESCRIPTION:
GL-ONC1, an oncolytic vaccinia virus, has shown the ability to preferentially locate, colonize and destroy tumor cells in more than 40 different human tumors. A First-in-Man, Phase I clinical study focusing on the safety and tolerability of GL-ONC1 intravenously administered to patients with a variety of advanced solid tumor entities has shown that GL-ONC1 is well-tolerated at therapeutic dose levels, with documented evidence of antitumor activity. Preclinical studies have further shown synergistic effects with the use of chemotherapy (Cisplatin) and viral therapy with GL-ONC, as well as favorable results when cancer cells are irradiated and then treated with GL-ONC1 in animal models. This Phase I study seeks to evaluate the safety, tolerability and early signs of efficacy of GL-ONC1 administered intravenously in combination with standard of care (SOC) radiation therapy (RT) and cisplatin (CDDP)in patients with locoregionally advanced head and neck cancer. Patients will be individually assessed for safety and dose limiting toxicity. Viral colonization in tumors, replication and anti-tumoral activity will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of histologically or cytologically documented Stage III to IVB primary, non-metastatic head and neck cancer for newly diagnosed patients with no prior disease-related treatment (e.g., chemotherapy, radiation treatment, surgery, etc.).
* American Joint Committee on Cancer (AJCC) Stage III-IVB disease (2010 manual, 7th edition), based on standard diagnostic workup.
* 18 years or older.
* ECOG performance status of ≤ 2.
* Laboratory data obtained within 14 days prior to Treatment Day 1, with adequate hepatic and renal function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3;
  * Platelets ≥ 100,000 cells/mm3;
  * Hemoglobin ≥ 8.0 g/dL;
  * Bilirubin ≤ 1.5 mg/dL;
  * AST or ALT ≤ 2× upper limit of normal (ULN);
  * Serum creatinine ≤ 1.5 mg/dL;
  * Creatinine clearance (CC) ≥ 50 mL/min.
* Pulse oximetry reading of 92% or higher at rest on room air.
* Signed informed consent
* Women of childbearing potential must have a negative serum pregnancy test and agree to practice effective birth control during treatment phase and up to 60 days after the last virus application.
* Male patients must agree to practice effective birth control during the study and for 60 days following administration of last treatment of virus.

Exclusion Criteria:

* Clinical, radiographic, or pathologic evidence of distant metastatic disease.
* Patients with fever, active immunosuppressive systemic infection or a suppressed immune system, including AIDS or HIV positivity and known hepatitis infections (HCV or HBC. Eligible patients must have an HIV test conducted within 4 weeks prior to study enrollment with a negative test result.
* Any form of prior anti-cancer treatment.
* Disease-related surgery, excluding biopsy.
* Patients with CNS (Central Nervous System) tumors.
* Any other open wounds.
* Concurrent small pox vaccination for 4 weeks before study therapy and during study treatment.
* Patients on immunosuppressive therapy or with immune system disorders, including autoimmune diseases.
* Prior splenectomy.
* Previous organ transplantation.
* Patients with clinically significant dermatological disorders, as judged by the clinical investigator (e.g., eczema or psoriasis), any skin lesions or ulcers, any history of atopic dermatitis, or any history of Darier's disease (Keratosis Follicularis).
* Clinically significant cardiac disease (New York Heart Association: Class III or IV).
* Dementia or altered mental status that would prohibit informed consent.
* Known allergy to ovalbumin or egg products.
* Prior gene therapy treatments or prior therapy with cytolytic virus of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by the number of patients with Adverse Events, as well as type of AE and frequency | Baseline up to week 23 Post-treatment
  Evaluation of changes in laboratory tests (hematological, chemistry), immunogenicity and physical examination

SECONDARY OUTCOMES:
Presence of Virus in Tumor | At baseline (Within 4 weeks of Treatment Day 1); 9-13 days post viral injection
  Analysis of tumor tissue (obtained through surgical or core biopsy if accessible from consenting patients) following viral treatment.
Determine Initial Susceptibility of tumor to viral infection | At baseline (Within 4 weeks of Treatment Day 1)
  Evaluate susceptibility of initial biopsied tumor to viral infection in cell cultures (for patients consenting to biopsy and where tumor is accessible).
Anti-Tumor Activity (Early Efficacy) | Change from baseline up to week 23 Post-treatment (week 23)
  Assessing changes in tumor measurement through physical examination, CT or CT/PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Loren K Mell, MD, Principal Investigator — Moores UC San Diego Cancer Center
Locations (1):
- Moores UC San Diego Cancer Center, La Jolla, California, United States